CLINICAL TRIAL: NCT04275232
Title: The Use of Allogenic Plasma Aliquots as a Source of Plasminogen in the Treatment of Ligneous Conjunctivitis, Clinical Trial of One Case
Brief Title: Allogenic Plasma Aliquots in the Treatment of Ligneous Conjunctivitis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Dorothy Bautista, MD (Other)
Collaborators: Canadian Blood Services (Other)
Responsible Party: Sponsor-Investigator, Dorothy Bautista, MD, Clinical Professor, Memorial University of Newfoundland
Organization: Memorial University of Newfoundland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DVB-LC-1
Record Dates: First submitted 2020-02-07; First posted 2020-02-19 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Ligneous Conjunctivitis, Left Eye
MeSH Terms: conditions — Plasminogen Deficiency, Type I

STUDY DESIGN:
Intervention Model Description: The patient will receive treatment with the interventional biologic product when she experiences recurrences of ligneous conjunctivitis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogenic Plasma Aliquots (Experimental): Allogenic Plasma Aliquots to be used as eye drops in the treatment of recurrences of ligneous conjunctivitis. Two drops will be administered to the affected eye, every 1 to 4 hours, depending on severity of the recurrence.
  Interventions: Biological: Allogenic plasma aliquots, a source of plasminogen

INTERVENTIONS:
Biological: Allogenic plasma aliquots, a source of plasminogen — Plasma eye drops, a source of plasminogen

SUMMARY:
Allogenic plasma aliquots, used as eye drops, will provide a source of plasminogen in the treatment of ligneous conjunctivitis. The investigational product will be available through written request from the Sponsor-Investigator to Canadian Blood Services, as approved by Health Canada.

DETAILED DESCRIPTION:
Ligneous conjunctivitis is a chronic progressive disorder of the conjunctival mucosa which occurs secondary to plasminogen deficiency. The condition is characterized by thick, fibrous pseudo membranes adherent to the conjunctival surface of the eye lid.The investigational product, allogenic plasma aliquots, is a source of plasminogen. It will be used as eye drops, to treat recurrences of these pseudo membranes by providing the plasminogen required for fibrinolysis. The allogenic plasma aliquots are prepared by Canadian Blood Services. An initial supply of 680 vials was made available through the Special Access program, upon approval by Health Canada. Through this Clinical Trial, additional allogenic plasma aliquots will be available when required to treat recurrences of the pseudo membranes. The study has been conditionally approved by local HREB, pending registration with clinicaltrials.gov

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed with ligneous conjunctivitis associated with Type 1 plasminogen deficiency

Exclusion Criteria:

* Subject has concurrent eye disease which prevents use of the investigational drug

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Clinical trial involves one patient (female)
Enrollment: 1 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Resolution of pseudo membrane associated with ligneous conjunctivitis | From date of first documented recurrence of pseudo membranes up to two years, starting from the date of enrolment
  Patient to be observed daily to every few weeks for resolution, based on clinical observation

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy V Bautista, MD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

REFERENCES:
- [Background] Kizilocak H, Ozdemir N, Dikme G, Koc B, Atabek AA, Cokugras H, Iskeleli G, Donmez-Demir B, Christiansen NM, Ziegler M, Ozdag H, Schuster V, Celkan T. Treatment of plasminogen deficiency patients with fresh frozen plasma. Pediatr Blood Cancer. 2018 Feb;65(2). doi: 10.1002/pbc.26779. Epub 2017 Sep 6. PMID 28876531
- [Background] Ku JY, Lichtinger A, Yeung SN, Kim P, Cserti-Gazdewich C, Slomovic AR. Topical fresh frozen plasma and heparin treatment of ligneous conjunctivitis in a Canadian hospital setting. Can J Ophthalmol. 2012 Oct;47(5):e27-8. doi: 10.1016/j.jcjo.2012.03.025. Epub 2012 Jul 13. No abstract available. PMID 23036559
- [Background] Pergantou H, Likaki D, Fotopoulou M, Katsarou O, Xafaki P, Platokouki H. Management of ligneous conjunctivitis in a child with plasminogen deficiency. Eur J Pediatr. 2011 Oct;170(10):1333-6. doi: 10.1007/s00431-011-1483-9. Epub 2011 May 31. PMID 21625933
- [Background] Ang MJ, Papageorgiou KI, Chang SH, Kohn J, Chokron Garneau H, Goldberg RA. Topical Plasminogen as Adjunctive Treatment in Recurrent Ligneous Conjunctivitis. Ophthalmic Plast Reconstr Surg. 2017 Mar/Apr;33(2):e37-e39. doi: 10.1097/IOP.0000000000000694. PMID 27065432
- [Background] Shapiro AD, Nakar C, Parker JM, Albert GR, Moran JE, Thibaudeau K, Thukral N, Hardesty BM, Laurin P, Sandset PM. Plasminogen replacement therapy for the treatment of children and adults with congenital plasminogen deficiency. Blood. 2018 Mar 22;131(12):1301-1310. doi: 10.1182/blood-2017-09-806729. Epub 2018 Jan 10. PMID 29321155
- [Background] Conforti FM, Di Felice G, Bernaschi P, Bartuli A, Bianco G, Simonetti A, Buzzonetti L, Valente P, Corsetti T. Novel plasminogen and hyaluronate sodium eye drop formulation for a patient with ligneous conjunctivitis. Am J Health Syst Pharm. 2016 Apr 15;73(8):556-61. doi: 10.2146/ajhp150395. PMID 27045067